CLINICAL TRIAL: NCT05015842
Title: Effectiveness of Kinesio Tapping for the Treatment of Patients With Acute Low Back Pain: A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NCS University System (Other)
Responsible Party: Principal Investigator, Hazrat Bilal PT, Assistant Professor, NCS University System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DIR/KMU-ASR&B/EK/000678
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Low Back Pain
Keywords: Low back pain, Kinesio tapping, conventional physical therapy, Oswestry disability index
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Tapping plus Conventional Physical Therapy - Experimental Group (Experimental): Both groups received conventional physical therapy treatment consisting of therapeutic exercise, heat therapy and manual therapy. All the patients received manual therapy techniques that including joint mobilization and therapeutic exercise that including piriformis stretching as well as bridging exercises to strengthen the core stability muscles (i.e., strengthening of transverses abdominis, erector spinae and lumbar multifidus).
  The KT was applied to the back once a week with a treatment duration of 2 weeks. Each KT was applied for continuous three days and the next KT was applied after a break of two days. Each participant in the experimental group was assessed for any allergy reaction of the skin to KT.
  Interventions: Other: Conventional Physical Therapy; Other: Kinesio Tapping
- Conventional Physical Therapy alone - Control Group (Other): Both groups received conventional physical therapy treatment consisting of therapeutic exercise, heat therapy and manual therapy. All the patients received manual therapy techniques that including joint mobilization and therapeutic exercise that including piriformis stretching as well as bridging exercises to strengthen the core stability muscles (i.e., strengthening of transverses abdominis, erector spinae and lumbar multifidus).
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Conventional Physical Therapy — This is a combine protocol of different therapeutic exercises and heat therapy.
Other: Kinesio Tapping — Kinesio Tapping is an adhesive and elastic fiber used for different outcomes like pain and swelling reduction among physical therapists.
  Arms: Kinesio Tapping plus Conventional Physical Therapy - Experimental Group

SUMMARY:
The objective of the study was to determine the effectiveness of Kinesio Taping (KT) for the treatment of patients with acute low back pain.

In this study a total of 56 patients with acute low back pain were randomly allocated to the experimental group, KT along with conventional Physical therapy (PT), or the control group, conventional PT alone.

DETAILED DESCRIPTION:
The objective of the study was to determine the effectiveness of Kinesio Taping (KT) for the treatment of patients with acute low back pain.

In this study a total of 56 patients with acute low back pain were randomly allocated to the experimental group, KT along with conventional Physical therapy (PT), or the control group, conventional PT alone. 28 Patients received KT in addition to conventional PT while 28 patients received conventional PT alone for two weeks. Oswestry disability index (ODI) and numeric pain rating scale (NPRS) were used for the measurement of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Both Genders
* Age between 18 and 60 years
* History of LBP less than

Exclusion Criteria:

* Patients having diagnosed conditions of spondylolisthesis, spondylosis, lumbar stenosis, spinal tumor, lumber fracture, renal disease and trauma were excluded from the study.
* Patients either with chronic LBP (duration more than 3 months) or contraindicated to KT (skin allergy or pre-existing skin lesion or infection) were also excluded.
* Female Pregnant patients were also excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  Pain was measured on numerical pain rating scale. it is a scale with score from 0 to 10 where 0 is no pain and 10 is maximum pain. The minimum score mean better outcome while higher score mean worse outcome. simply lesser the score better would be the outcome.

SECONDARY OUTCOMES:
Functional Disability | 2 weeks
  Functional disability was measured using Oswestry Disability Index (ODI. ODI score was converted to percentage so the score ranges from 0% to 100%. Where 0% mean no disability and 100 mean very severe (maximum) disability. The minimum score mean better outcome while higher score mean worse outcome. simply lesser the score better would be the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Haider Darain, PhD, Study Director — Khyber Medical University
Locations (1):
- NCS University System, Department of Physical Therapy and Rehabilitation, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No